CLINICAL TRIAL: NCT07065253
Title: CHOICE KERGUELEN 1: Consequences of Longterm Confinement on Immunity in the Sub-Antarctic Islands: Inclusion of Volunteers Before Departure to the Kerguelen Islands
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Institut Polaire Français Paul-Emile Victor (IPEV) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 49RC25-0245
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Human Health in Extreme Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, PBMCs, plasma, serum, urine, saliva, stools, hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HD (healthy donors)
  Interventions: Other: blood ponction; Other: urines collection; Other: hair collection; Other: saliva collection; Other: stools collection

INTERVENTIONS:
Other: blood ponction — blood ponction
Other: urines collection — urines collection
Other: hair collection — hair collection
Other: saliva collection — saliva collection
Other: stools collection — stools collection

SUMMARY:
Living for long periods in extreme environments-like Antarctic research stations or space missions-can have a significant impact on human health, especially on the immune system. Scientists have observed that people in such isolated conditions often experience more infections and a reactivation of viruses that usually stay dormant in the body, such as Herpes viruses. These changes affect both parts of the immune system: the rapid-response "innate" system and the slower, more specific "adaptive" system.

These immune disruptions may be caused by multiple stressors: ongoing psychological stress, disturbed sleep and light cycles (circadian rhythm disruption), and the challenges of living in confined, isolated, and extreme environments. While space missions and Antarctic overwintering programs have provided some insight into these issues, scientists still lack a detailed understanding of how the immune system adapts-or fails to adapt-over time in such conditions.

To help fill this gap, the CHOICE Kerguelen 1 study will recrut a group of healthy young adults who will spend one year (from November 2025 to November 2026) in Port-aux-Français, a remote French research station on the Kerguelen Islands in the sub-Antarctic. These volunteers are participating in a civic service program and will be living in a highly isolated environment for the duration of their mission. The CHOICE Kerguelen 1 study is conducted in collaboration with the French Polar Institute (IPEV).The goal of the study is to collect and store a broad range of biological samples-including blood, saliva, stool, urine, and hair-from these volunteers before they leave for the island, to have baseline medical state and baseline biological samples. These samples will integrate in to healthy volunteer biobank of CHU Angers, a type of biological archive that provided control samples for CHOICE Kerguelen 2 - a clinical study relating to follow-up of volunteers during civic service on the Kerguelen Islands

ELIGIBILITY:
Inclusion Criteria :

* healthy people aged > 18 years
* Participant affiliated with or benefiting from a social security system
* Participant has signed informed consent
* Participant staying as an overwintering member at Kerguelen from November 2025 to November 2026

Exclusion Criteria:

* age < 18 years
* Pregnant, breastfeeding, or postpartum woman
* immunocompromised people (primary immunodeficiency, HIV infection or immunosupressive treatment)
* Person refusing to participate in the study
* Person with a history of autoimmune disease - -Person deprived of liberty by judicial or administrative decision
* Person undergoing involuntary psychiatric treatment
* Person subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French civic service volunteer
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Blood samples | At inclusion (before overwintering)
  Blood samples
Saliva samples | At inclusion (before overwintering)
  Saliva samples
Urine samples. | At inclusion (before overwintering)
  morning urine samples.
Hair samples | At inclusion (before overwintering)
  Hair samples
Stool samples | At inclusion (before overwintering)
  Stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Charline MIOT, Principal Investigator — University Hospital, Angers
Locations (1):
- Paul Emile Victor Polar Institute, Plouzané, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).